CLINICAL TRIAL: NCT00469365
Title: A Randomized Controlled Trial of Two Pharmacy Interventions to Improve Refill Adherence for Chronic Disease Medications
Brief Title: Pharmacy Interventions to Improve Chronic Disease Medication Refill
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P01HS010871 (AHRQ)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes; Hypertension; Hyperlipidemia; Heart Diseases; Depression; Psychoses
Keywords: clinical trial, medication adherence, pharmacy intervention; Patients with specific chronic diseases
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias; Heart Diseases; Depression; Psychotic Disorders; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: pharmacist contact with the patient via telephone
Behavioral: Pharmacist contact with the patient's physician via fax
Behavioral: Usual care

SUMMARY:
Compare the effectiveness of 3 strategies by pharmacists to decrease the time to refill of prescriptions for common chronic diseases (diabetes, hypertension, hyperlipidemia, heart failure, depression, psychoses).

DETAILED DESCRIPTION:
The design was a multi-site 8-month randomized, controlled clinical trial with the patient as the unit of randomization. The Institutional Review Board at the Medical University of South Carolina approved the study. The setting included 9 pharmacies within a medium-sized grocery store chain in South Carolina. The 9 pharmacies were selected to ensure an adequate sample size and sufficient representation by patients with respect to geographic region (urban, suburban, and rural), race/ethnicity, and socioeconomic background. Individual pharmacy staff were informed by their district manager (P.P.) that they were required to participate in the project. Beginning January 16, 2006 and continuing through August 29, 2006, all patients who were at least 7 days overdue for a qualified prescription were identified on a weekly basis (i.e. every Monday morning) using the centralized computer database. Patients identified as being overdue for a qualified medication were assigned a unique study identification number and randomized using a simple randomization technique operationalized within a Microsoft® Access® database. The randomization was based on a permuted block design with a block size of 3, with each patient thus having a one-third chance of being placed in any one of the 3 treatment arms.After eligible patients were identified and randomized each week, there were 3 different protocols followed, depending on the assigned treatment arm. The 3 treatment arms included 1) pharmacist contact with the patient via telephone, 2) pharmacist contact with the prescribing physician via facsimile, and 3) usual care.There were a total of 3,048 patients into arms 1 (n=1018), 2 (n=1016), and 3 (n= 1014). The study was designed to detect relatively small differences in the outcomes of interest. Baseline comparisons across treatment arms in the characteristics of patients and medications were made using t-tests and chi-square tests, as appropriate. For the analyses of study outcomes, an intent-to-treat approach was used. Statistical models were constructed to compare outcomes among the 3 treatment arms, after first examining whether significant interaction between treatment arm and medication disease classification was present. For the analyses of secondary outcomes, all of which were binary in nature, multivariable logistic regression models were used, with treatment arm as the key independent variable of interest, adjusting for the same covariates used in the primary analyses.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were at least 7 days overdue for a qualified prescription were identified on a weekly basis (i.e. every Monday morning) using the centralized computer database. A qualified prescription was defined as having at least 2 refills remaining, a duration of at least a 30 days' supply, and having been written for any one of a number of chronic disease medications identified by a clinical pharmacist (A.M.W.). The medications of interest were those indicated for chronic treatment of diabetes mellitus, hypertension, hyperlipidemia, heart failure, depression, and psychoses. Medications that treat any combination of the specified diseases were allowed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3048 (Actual)
Dates: Start 2006-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the number of days from the index date until the next date on which the patient filled a prescription for any qualified medication, or until the end of the study follow-up period.

SECONDARY OUTCOMES:
Secondary outcomes included indicators for whether the patient filled any medication within 30 days for their chronic disease, and whether the patient filled any medication within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Nietert, PhD, Principal Investigator — Medical University of South Carolina; Barbara C Tilley, PhD, Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States